CLINICAL TRIAL: NCT04863950
Title: A Phase II, Investigator-Initiated Study of Imipramine Hydrochloride and Lomustine in Recurrent Glioblastoma
Brief Title: Investigator-Initiated Study of Imipramine Hydrochloride and Lomustine in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, William Kelly, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 20-0148
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine; Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Imipramine Hydrochloride/Lomustine (Experimental)
  Interventions: Drug: Lomustine; Drug: Imipramine Hydrochloride

INTERVENTIONS:
Drug: Lomustine — For surgical cohort patients, lomustine will be initiated (C1D1) within 6 weeks of surgery as soon as patient is deemed by the investigator (or designee) to be recovered enough for chemotherapy. Initiation of lomustine must be initiated within 6 weeks. If patient cannot be safely initiated on lomustine within this timeframe then they will be replaced.
  For non-surgical cohort patients (the decision for surgery is made independent of study participation), lomustine will be initiated on C1D1.
  For both cohorts, lomustine will be administered as 110 mg/m2 PO once every 6 weeks.
  Other Names: Gleostine
Drug: Imipramine Hydrochloride — For the surgical cohort, imipramine hydrochloride will be initiated within a minimum of 16 days to a maximum of 3 weeks prior to surgery. Imipramine hydrochloride will be administered as 50mg PO (oral) QHS (at bedtime) for 4 days followed by a dose increase (taper-up) of 50mg/day every fourth day to attain a maximum dose of 200mg/day in 16 days.
  For non-surgical cohort patients (the decision for surgery is made independent of study participation), imipramine hydrochloride will be initiated on Cycle 1 Day 1. Imipramine hydrochloride will be administered as 50mg PO (oral) QHS (at bedtime) for 4 days followed by a dose increase (taper-up) of 50mg/day every fourth day, if tolerated, to attain a maximum dose of 200mg/day in 16 days.
  Other Names: Trofranil

SUMMARY:
This study is designed as a single center, prospective, open label, single-arm therapeutic trial with both surgical and non-surgical cohorts.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age
* The subject has the ability to understand the purposes and risks of the study and to have signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* The subject has histologically confirmed glioblastoma
* The subject has progression following standard combined modality treatment with radiation and temozolomide chemotherapy
* The subject has an ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* The subject has a life expectancy of at least 3 months
* The subject has acceptable liver function:
* Bilirubin ≤ 1.5 times upper limit of normal
* AST (aspartate aminotransferase) (SGOT) and ALT (alanine transaminase 0 (SGPT) ≤ 3.0 times upper limit of normal (ULN)
* The subject has acceptable renal function:
* Serum creatinine ≤ULN
* The subject has acceptable hematologic status (without hematologic support):
* ANC (absolute neutrophil count) ≥1500 cells/uL
* Platelet count ≥100,000/uL
* Hemoglobin ≥9.0 g/dL
* All women of childbearing potential (not surgically sterilized or at least 1 year post-menopausal) must have a negative serum pregnancy test. Additionally, male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.

Exclusion Criteria:

* The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug.
* The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.
* The subject is unable to undergo MRI scan (eg, has pacemaker).
* The subject has received enzyme-inducing anti-epileptic agents within 14 days of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone).
* The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≤ 1 from AEs (except alopecia, anemia and lymphopenia) due to surgery, antineoplastic agents, investigational drugs, or other medications that were administered prior to study drug.
* The subject has evidence of wound dehiscence.
* The subject is pregnant or breast-feeding.
* The subject has a history of cardiac disease, including arrhythmia, conduction abnormality, congenital prolonged QT syndrome, myocardial infarction, unstable angina pectoris or congestive heart failure.
* A prolonged QTc rhythm noted during initial ECG >480 ms.
* The subject has serious intercurrent illness, such as:
* Hypertension (two or more blood pressure [BP] readings performed at screening of > 150 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment

  * Non-healing wound, ulcer, or bone fracture
  * Untreated hypothyroidism
  * Unhealed rectal or peri-rectal abscess
  * Uncontrolled active infection
  * Stroke, or transient ischemic attack within 6 months
* The subject has received any of the following prior anticancer therapy:

  * Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy (RIT), or intra-operative radiotherapy (IORT). Note: stereotactic radiosurgery (SRS) is allowed
  * Non-bevacizumab systemic therapy (including investigational agents and small- molecule kinase inhibitors) or non-cytotoxic hormonal therapy (eg, tamoxifen) within 7 days or 5 half-lives, whichever is shorter, prior to first dose of study drug
  * Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
  * Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to first dose of study drug
  * Prior treatment with carmustine wafers
* Any current psychosis, uncontrolled mood disorder (as assessed by investigator) or suicidal ideation. Additionally, current or history of bipolar disorder is excluded.
* Patients currently using SSRI, SNRI, MAO inhibitors, tramadol or trazodone who are unwilling to undergo taper.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William Kelly, MD, Principal Investigator — The University of Texas Health Science Center - Mays Cancer Center
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided